CLINICAL TRIAL: NCT06546800
Title: SPECIAL INVESTIGATION FOR ABRYSVO INTRAMUSCULAR INJECTION -INVESTIGATION IN INDIVIDUALS AGED 60 YEARS OR OLDER-
Brief Title: SPECIAL INVESTIGATION FOR ABRYSVO IN INDIVIDUALS AGED 60 YEARS OR OLDER
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3671019
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: Respiratory syncytial virus infection; RSV Vaccine; Individuals aged 60 years or older; Post Marketing Study
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — abrysvo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- RSVpreF vaccine: Individuals aged 60 years or older who has been vaccinated with Abrysvo for the first time.
  Interventions: Biological: RSVpreF vaccine

INTERVENTIONS:
Biological: RSVpreF vaccine — Injection in the muscle, 1 dose 0.5mL
  Other Names: Abrysvo

SUMMARY:
This post-marketing study is a multicenter cohort study in individuals aged 60 years or older vaccinated with Abrysvo (RSV vaccine）designed to confirm the safety in individuals aged 60 years or older under actual clinical practice in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 60 years or older who have been vaccinated with Abrysvo for the first time after Abrysvo is launched. Those who have previously participated in the clinical trials of this product will be excluded.
2. Vaccinated participants (or his/her legally acceptable representative) who understand the information on this study and have provided written consent regarding their participation in the study.

Exclusion Criteria:

-There are no exclusion criteria for this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 60 years or older who have been vaccinated with Abrysvo for the first time.
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of individuals aged 60 years or older reporting Adverse Reactions for 28 days after vaccination. | From the day of vaccination up to 28 days after vaccination.
  Adverse reaction (including serious) in individuals aged 60 years or older will be assessed.
Percentage of individuals aged 60 years or older reporting Serious Adverse Reactions from the day of vaccination up to 28 days after vaccination. | From the day of vaccination up to 28 days after vaccination.
  Serious adverse reaction in individuals aged 60 years or older will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671019